CLINICAL TRIAL: NCT02063490
Title: A Nurse-led Multifactorial Intervention to Improve Phosphate Binder Adherence: Results From a One-year Clinical Trial
Brief Title: Nurse-led Intervention to Improve Phosphate Binder Adherence
Acronym: MedAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiteit Antwerpen (Other)
Responsible Party: Principal Investigator, Yoleen Van Camp, Dra., Universiteit Antwerpen
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UA-B300201111744
Record Dates: First submitted 2014-02-10; First posted 2014-02-14 (Estimated); Last update posted 2014-02-14 (Estimated); Status verified 2014-02

CONDITIONS: End Stage Renal Failure on Dialysis
Keywords: Adherence; dialysis; intervention; nurse-led; phosphate binders; trial

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Adherence support (Experimental): One-time preparatory intervention offering adherence prerequisites (knowledge, social support and skills)
  + One-year monthly individualised counselling sessions with a standardised intervention sheet listing the most prevalent problems with possible solutions
  Interventions: Behavioral: Adherence support
- Control arm (No Intervention): Standard care

INTERVENTIONS:
Behavioral: Adherence support — One-time preparatory intervention offering adherence prerequisites (knowledge, social support and skills)
  + One-year monthly individualised counselling sessions with a standardised intervention sheet listing the most prevalent problems with possible solutions
  Other Names: Nurse-led multifactorial intervention; Individualised management
  Arms: Adherence support

SUMMARY:
The study aim is to test the efficacy of one-year nurse-led interventions to improve the medication intake behaviour of chronic dialysis patients. The investigators hypothesis is the interventions leading to a 15% mean increase in intake, compared to standard care.

DETAILED DESCRIPTION:
Background Phosphate binder nonadherence is ubiquitous. The results of adherence enhancing interventions are often disappointing. The aim is to test a nurse-led multifactorial intervention to enhance phosphate binder adherence.

Methods In a quasi-experimental clinical trial, phosphate binder adherence was measured electronically in 135 hemodialysis patients for one year and phosphatemia measured monthly. For all patients, months 1-2 were baseline (no interventions were performed). The intervention arm was given 1 "preparatory" intervention and then monthly 8 "maintenance" individualized management sessions. The control arm received standard of care.

ELIGIBILITY:
Inclusion Criteria:

* adult (≥18)
* chronic hemodialysis ≥1 month
* treated with phosphate binders
* Dutch-speaking

Exclusion Criteria:

* receiving professional medication care
* cognitive impairment
* nursing home residents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2011-11; Primary Completion 2012-11 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Medication adherence | One year
  The intake of medication (phosphate binders) was monitored continuously for one year through electronic monitoring with the Medication Event Monitoring System (MEMS). Medication containers are filled with patients' phosphate binders and then capped with MEMS-caps registering the time and date of each opening and thus presumed intake of the medication in the box.
  Mean adherence was calculated as the proportion of prescribed doses taken, averaged per month (e.g. patients with a ter in die regimen (84 doses/month) and taking them all 84 would have a mean adherence of 84/84=100%). Nonadherence was defined as a mean adherence <80%.

SECONDARY OUTCOMES:
Serum phosphate | Monthly for one year
  Serum phosphate was gathered monthly from patients' charts. In addition to mean serum phosphate per month we dichtomised this outcome measure with >5mg/dL representing uncontrolled phosphatemia.
Patient knowledge | At study start and end (after one year)
  Knowledge was measured by ten multiple-choice questions about the phosphate cycle, phosphate binder pharmacodynamics and dietary recommendations, developed in previous research and added as appendix in a previous article (Van Camp Y, Vrijens B, Abraham I, et al. Adherence to phosphate binders in hemodialysis patients: prevalence and determinants. J Nephrol 2013; JNEPHROL-D-13-00176R1: Publicatin in process)
Social support | At study start and end (after one year)
  Social support was measured by eleven questions assessing perceived support in general and support with taking phosphate binders specifically, developed in previous research and added as appendix in a previous article (Van Camp Y, Vrijens B, Abraham I, et al. Adherence to phosphate binders in hemodialysis patients: prevalence and determinants. J Nephrol 2013; JNEPHROL-D-13-00176R1: publication in process)

CONTACTS AND LOCATIONS:
Overall Officials: Yoleen PM Van Camp, MScN, Principal Investigator — Universiteit Antwerpen
Locations (3):
- Belgium (3):
  - Dialysis hospital unit 1, Antwerp
  - Dialysis hospital unit 3, Antwerp
  - Dialysis hospital unit 2, Turnhout